CLINICAL TRIAL: NCT02344849
Title: An Open, Single-center, Phase 1 Study to Evaluate Safety of Autologous Bone Marrow Derived Mesenchymal Stem Cell in Erectile Dysfunction.
Brief Title: Safety of Autologous Bone Marrow Derived Mesenchymal Stem Cells in Erectile Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cellgram-ED
Record Dates: First submitted 2015-01-13; First posted 2015-01-26 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesenchymal stem cell (Experimental): Patients will receive single intracavernous injection of Mesenchymal stem cell. Oral PDE5-inhibitor can take on demand.
  Interventions: Drug: mesenchymal stem cell

INTERVENTIONS:
Drug: mesenchymal stem cell — Patients will receive single injection of Cellgram-ED( 30,000,000 mesenchymal stem cell) intracavernously.
  Other Names: Cellgram-ED

SUMMARY:
This phase I clinical trial is designed to evaluate the safety of autologous Mesenchymal Stem Cells (MSC) injected intracavernously.

DETAILED DESCRIPTION:
Cellgram-ED is autologous bone marrow-derived mesenchymal stem cells ex vivo expanded for approximately 30 days. Ten patients (Diabetes -associated ED; 5 patients, Postprostatectomy; 5patients) will be injected Cellgram-ED directly into the intracavernous. Patient will be evaluated the safety and potential efficacy of MSC.

ELIGIBILITY:
Inclusion Criteria:

Postprostatectomy Erectile Dysfunction

* A man aged 20 or older
* Who is willing to consent to participate in the study concerned with improving sexual activity after prostatectomy, the man has maintained normal sexual activity prior to prostatectomy
* Prior to prostatectomy PSA (prostate specific antigen) level<10 ng/mL
* At the time of Prostatectomy, Pathological Gleason sum ≤7
* At the time of Prostatectomy, Pathological stage ≤ T2c
* 2 years or more postprostatectomy patients with PSA level ≤ 0.04 ng/mL without additional therapy after prostatectomy
* Who cannot satisfy sexual activity(more than 4 times) with proper sexual stimulation in spite of taking maximum dose of oral PDE5I(phos-phodiesterasetype-5 inhibitors) within last 8weeks.
* IIEF, EF(erectile function) domain score is under 17
* Have a consistent partner who is willing to engage in sexual activity more than twice per month during the study.

Diabetes-associated Erectile Dysfunction

* HbA1c is between 6.5% and 10% of man over 20 years of age with diabetes
* Who cannot satisfy sexual activity(more than 4 times) with proper sexual stimulation in spite of taking maximum dose of oral PDE5I within last 8weeks.
* IIEF, EF domain score is under 17
* Who is willing to consent to participate in the study concerned with improving sexual activity
* Have a consistent partner who is willing to engage in sexual activity more than twice per month during the study.

Exclusion Criteria:

* History of bone marrow disorders
* Serum AST/ALT > 3 X upper limit of normal or Creatinine > 1.5 X upper limit of normal
* History of hypersensitivity against a gentamycin
* Severe cardiovascular disease(angina, arrhythmia, cardiac failure, stroke), kidney failure, respiratory failure
* Positive for human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) and syphilis test
* Positive for PSA or CEA or AFP (Carcinoembryonic antigen), history of cancer in the last five years (except Prostatic cancer) Uncontrolled hypertension or hypotension (systolic blood pressure > 170 or < 90 mm Hg, diastolic pressure > 100 or < 50 mm Hg)
* HbA1c exhibit greater than 10%
* Men on anticoagulant treatment
* Have a severe infectious disease
* Testosterone level is less than 200ng/dl
* Have a penile implant or willing to it
* Patients with morphological changes of the penis
* Patient's partner is trying to conceive during the trial period
* Unwilling to participate in the study
* Participating in other clinical trials in the past 30 days
* Unable to compliance with protocol
* Inappropriate patients to participate in the study according to the investigator

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07; Primary Completion 2018-01-31 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events | 12month
  Analyze the laboratory, vital sign, physical exam results from baseline to end of the study for investigate adverse reactions and view safety.
  An SAE suggests a significant hazard, contraindication, side-effect, or precaution. With respect to human clinical experience, this includes any event that:
  Results in death. Is life-threatening.* Requires in-patient hospitalization or prolongation of existing hospitalization.
  Results in persistent or significant disability/incapacity. Is a congenital anomaly/birth defect. Other medically important condition
  Life-threatening in the definition of a SAE or adverse reaction refers to an event in which the patient was at risk of death at the time of event; it does not refer to an event, which hypothetically might have caused death if it were more severe.

SECONDARY OUTCOMES:
Change From Baseline in the International Index of Erectile Function(IIEF) | month 1, 3, 6, 9 and 12
  Description of the average variation from the screening value in each group using the Student's preordered t-test (Wilcoxon's signed bank test).
  Function domain
  * Erectile Function (Q1,2,3,4,5,15) : Min 6 ~ Max 30
  * Orgasmic Function (Q9,10) : Min 2 ~ Max 10
  * Sexual Desire (Q11,12) : : Min 2 ~ Max 10
  * Intercourse Satisfaction (Q6,7,8): : Min 3 ~ Max 15
  * Overall Satisfaction (Q13,14) : Min 2 ~ Max 10
Penile Doppler Sonography, PDS | month 6, 12
  Change From Baseline in Peak systolic velocity (PSV) and End diastolic velocity (EDV), Evaluate Erection rigidity During the test.
  The normal maximum systolic blood flow of the cavernosal artery after injection of vasodilators is 30 cm / s or more.
  1. PDS results are obtained 5 min, 10 min, 15 min, 20 min, 25 min and 30 min after intracavernosal injection.
  2. The peak systolic velocity (PSV) is assessed as follows:
     >25 cm/s is considered to be normal, 20-25 cm/s is considered to be mild ED, 12-20 cm/s is considered to be moderate ED, <12 cm/s is considered to be severe arteriogenic impotence.
  3. The end diastolic velocity (EDV) is assessed as follows:
     * 5 cm/s is considered to be a normal value, >5 cm/s is considered to indicate a veno-occlusive disorder.
Change From Baseline in Sexual Encounter Profile (SEP) Question 2 | month 1, 3, 6, 9 and 12
  The SEP2 survey describes cumulative success rates for 30 days, 3 months, 6 months, 9 months and 12 months after cell treatment.
  SEP 2 Were you able to insert your penis into your partner's vagina? Yes or No SEP 3 Did your erection last long enough to have successful intercourse? Yes or No
Global Assessment Question (GAQ) | month 1, 3, 6, 9 and 12
  The GAQ survey describes cumulative success rates for 30 days, 3 months, 6 months, 9 months and 12 months after cell treatment.
  GAQ
  1. Did Cellgram-ED improve your Erectile Function? Yes or No
  2. If so, did Cellgram-ED improve the ability to have sex? Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Chungsu Kim, Ph.D, Principal Investigator — AIDS Malignancy Consortium
Locations (1):
- Asan medical center, Seoul, South Korea

REFERENCES:
- [Derived] You D, Jang MJ, Song G, Shin HC, Suh N, Kim YM, Ahn TY, Kim CS. Safety of autologous bone marrow-derived mesenchymal stem cells in erectile dysfunction: an open-label phase 1 clinical trial. Cytotherapy. 2021 Oct;23(10):931-938. doi: 10.1016/j.jcyt.2021.06.001. Epub 2021 Jul 27. PMID 34326007